CLINICAL TRIAL: NCT02924870
Title: Long-term Effect of an Health Education Program on Daily Physical Activity in Patients With Moderate to Very Severe Chronic Obstructive Pulmonary Disease
Acronym: EA-EPOC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Francisco Garcia-Rio, MD, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULP PI-4447
Record Dates: First submitted 2016-10-02; First posted 2016-10-05 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: health education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Conventional management. Treatment and follow-up according to conventional clinical practice (GesEPOC guidelines), including recommendations on healthy habits and lifestyle.
  Interventions: Other: Conventional management
- Intervention group (Experimental): Conventional management plus health education program. In addition to conventional treatment and follow-up, the patients will be referred to a nursing consultation for perform two health education sessions, at 15 and 30 days after hospital discharge.
  Interventions: Other: Health education program; Other: Conventional management

INTERVENTIONS:
Other: Health education program — 2 sessions, at 15 and 30 days after hospital discharge. The first session will consist of four stages:
  * Basic formation: basic lung anatomy and physiology, COPD concept, importance of tobacco, diagnostic tests for COPD, and how COPD is treated.
  * Care in COPD: diet, breathing exercises, physical exercise (walking, cycle, treadmill ...), lifestyle (clothing, hygiene, preening, exercise, rest, sexuality, social relations).
  * Management of conventional treatment: inhalers, oxygen therapy and smoking cessation.
  * Action Plan: the patient and the nurse will establish a target about the activities that the patient must perform as well as their frequency and duration, according to WHO guidelines.
  Second session: changes from the previous session; compliance with the physical activity plan and the deviation causes; weaknesses of the patient; skills in the management of inhalers, oxygen, and breathing exercises; and a new physical activity plan.
  Arms: Intervention group
Other: Conventional management — Treatment and follow-up according to conventional clinical practice (GesEPOC guidelines), including recommendations on healthy habits and lifestyle.

SUMMARY:
Main objective: To compare the level of physical activity (PAL) at 12 months in patients with moderate to very severe chronic obstructive pulmonary disease (COPD) between those who completed a health education program and those who did not.

Study patients. Subjects older than 35 years; diagnosis of moderate to very severe COPD (FEV1 <80% predicted), established at least 3 months; current or former smoker with an accumulated consumption >10 packs x year; and hospital admission for COPD exacerbation.

Design. Randomized, parallel and open-label clinical trial, controlled with conventional treatment.

Intervention: During hospitalization, selected patients will receive conventional treatment. At discharge, they will be randomized (1:1) to control group [treatment and follow-up according to conventional clinical practice] or intervention group [in addition to conventional treatment and follow-up, the patients will be referred to a nursing consultation for perform two health education sessions, at 15 and 30 days after hospital discharge].

Measurements. At 15 days and 12 months after discharge, the following determinations will be made: anthropometric characteristics; clinical evaluation (smoking history, date of COPD diagnosis, comorbidities, current medication; health care utilization; moderate or severe COPD exacerbations); questionnaires (mMRC, Charlson, COPD-specific co-morbidity test (COTE), COPD Assessment Test (CAT) and LCADL), spirometry and six-minutes walking test; and evaluation of daily physical activity using an accelerometer.

DETAILED DESCRIPTION:
Objectives: To compare the level of physical activity (PAL) at 12 months in patients with moderate-very severe COPD between those who completed a health education program and those who did not.

Secondary objectives: 1) To compare the average of steps per day at 12 months in patients with moderate-very severe COPD between the intervention group (conventional treatment plus health education program) and the control group (conventional treatment); 2) to compare the daily minutes of moderate to high intensity at 12 months between the intervention and control groups; 3) to compare the daily energy expenditure higher than 3 metabolic equivalents (METs) at 12 months between the intervention and control groups; 4) to compare the distribution profile of the daily physical activity (very sedentary, sedentary, moderately active) at 12 months between the intervention and control groups; 5) to evaluate the long-term effect of the health education program on the health-related quality of life of patients with moderate to very severe COPD; 6) to analyze the effect of the health education program on the risk and powered rate of moderate or severe COPD exacerbations; 7) to assess the relationship between the change of the PAL and the modification of the health-related quality of life and the number of moderate or severe exacerbations; and 8) to identify the determinants of a clinically relevant increase of the PAL (> 0.14 units) in patients with moderate to very severe COPD.

METHODS I. Study subjects. Patient selection will be held consecutively in the Department of Pneumology, University Hospital La Paz-Cantoblanco-Carlos III, according to the following criteria.

* Inclusion criteria: subjects older than 35 years; diagnosis of moderate to very severe COPD (FEV1 <80% predicted), according to the GesEPOC criteria [Arch Bronconeumol 2012;48 (Suppl 1):2-58], established at least 3 months; current or former smoker with an accumulated consumption >10 packs x year; and hospital admission for COPD exacerbation.
* Exclusion criteria: osteoarticular, neuromuscular or cognitive limitation that prevents ambulation; previous diagnosis of active neoplastic disease; institutionalized patients; alcohol consumption >60 g/day; patient belonging to another health sector in the Community of Madrid or other community; participation in another study within 6 months prior.

All participants must sign informed consent approved by the Ethics Committee of University Hospital La Paz.

II. Design. Randomized, parallel and open-label clinical trial, controlled with conventional treatment.

A. Protocol and intervention. During hospitalization, selected patients will receive conventional treatment. At discharge, they will be randomized (1:1) to:

* Control group. Treatment and follow-up according to conventional clinical practice (GesEPOC guidelines), including recommendations on healthy habits and lifestyle.
* Intervention group. In addition to conventional treatment and follow-up, the patients will be referred to a nursing consultation for perform two health education sessions, at 15 and 30 days after hospital discharge.

The first session will last about 90 minutes and will consist of four stages:

* Basic formation. The manual "Controlling the COPD", published by the Spanish Society of Pneumology and Thoracic Surgery (SEPAR) will be handed to participants. The nurse will individually review the following aspects: basic lung anatomy and physiology, COPD concept, importance of tobacco, diagnostic tests for COPD (spirometry, blood gases, sputum cultures, simple radiology, laboratory, walking test), and how COPD is treated.
* Care in COPD: diet, breathing exercises, physical exercise (walking, cycle, treadmill ...), lifestyle (clothing, hygiene, preening, exercise, rest, sexuality, social relations).
* Management of conventional treatment: inhalers, oxygen therapy and medications; integration of treatment, and adhesion; smoking cessation.
* Action Plan: the patient and the nurse will establish a target about the activities that the patient must perform as well as their frequency and duration, according to WHO guidelines.

The second session will last approximately 15 minutes and it will be scheduled a month later. Current situation of the patient and the changes from the previous session will be assessed; compliance with the physical activity plan and the deviation causes will be analyzed; the weaknesses of the patient will be strengthened (training, incentives); skills in the management of inhalers, oxygen, and breathing exercises will be tested; and a new physical activity plan will be maintained or intensified (WHO guidelines).

There are no therapeutic restrictions for the patients included in the study, which will be treated by their usual pulmonologist and other health professionals according to their clinical judgment. Therefore, no limitation is posed to change the usual treatment (including the prescription of oxygen therapy or noninvasive ventilation) or to schedule follow-up visits performed by the regular doctor.

B. Sample size. Considering a mean PAL value of 1.55 ± 0.265 in patients with moderate-severe COPD and an increase of 0.14 units as clinically relevant, since it is associated with a mortality reduction [Chest 2011;140:331-42], to detect a difference ≥0.14 units, by contrast bilateral hypothesis (with alpha risk=0.05, beta risk=0.20 and drop-out rate=10%), it is estimated to will be necessary to randomize 64 patients to each treatment arm.

III. Measurements. At 15 days and 12 months after discharge, the following determinations will be made:

1. Anthropometric characteristics (sex, age, weight, height, BMI and BSA).
2. Clinical evaluation: Smoking history (cigarettes/day, packs-year), date of COPD diagnosis, comorbidities, current medication; visits to primary care physician or pulmonologist (scheduled and unscheduled) and emergency room (date and cause), hospitalizations (date and cause) and periods off work (date and cause); number and date of moderate (prescription of antibiotics or systemic corticosteroids) or severe (hospitalization or stay in the emergency department >24 hours) exacerbations.
3. Questionnaires: mMRC dyspnea scale, Charlson and COTE comorbidity indices, CAT and LCADL.
4. Spirometry and six-minutes walking test, according current guidelines [Arch Bronconeumol 2013; 49: 388-401; Am J Respir Crit Care Med 2002; 166: 111-7].
5. Evaluation of daily physical activity. It will be made using a Sense Wear accelerometer (Body Media), that it will be placed on the no dominant arm for 7 consecutive days. The physical activity level (PAL) will be recorded. Depending on this parameter, the subjects will be classified as very sedentary (PAL <1.40), sedentary (PAL 1.40 to 1.69) or moderately active (PAL> 1.70). The mean of steps per day, minutes per day of moderate to high intensity (>3 METs) and daily energy expenditure >3 METs will be also determined.

IV. Statistical analysis. T-Student, Mann-Whitney and chi-square test for between-groups comparisons. Relationship analysis using Pearson correlation and multivariate regression models. Intention-to-treat evaluation of the main objective with imputation of missing data by a regression model. The effect of the intervention will be evaluated by the difference of change for each variable between the two groups using general linear models. The crude effect (only adjusted for baseline values) and the adjusted effect for several confounders (sex, age, BMI, smoking, treatment and FEV1%) will be determined.

ELIGIBILITY:
Inclusion Criteria:

* subjects older than 35 years
* diagnosis of moderate to very severe COPD (FEV1 <80% predicted), according to the GesEPOC criteria, established at least 3 months
* current or former smoker with an accumulated consumption >10 packs x year
* hospital admission for COPD exacerbation

Exclusion Criteria:

* osteoarticular, neuromuscular or cognitive limitation that prevents ambulation
* previous diagnosis of active neoplastic disease
* institutionalized patients; alcohol consumption >60 g/day
* patient belonging to another health sector in the Community of Madrid or other community
* participation in another study within 6 months prior.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Physical activity level | 12 months
  To compare the physical activity level at 12 months in patients with moderate-very severe COPD between the intervention group (conventional treatment plus health education program) and the control group (conventional treatment)

SECONDARY OUTCOMES:
Steps per day | 12 months
  To compare the average of steps per day at 12 months in patients with moderate-very severe COPD between the intervention group (conventional treatment plus health education program) and the control group (conventional management)
Daily minutes of moderate-high intensity activity | 12 months
  To compare the daily minutes of moderate to high intensity at 12 months between the intervention and control groups
Daily energy expenditure higher than 3 METs | 12 months
  To compare the daily energy expenditure higher than 3 METs at 12 months between the intervention and control groups
Profile of the daily physical activity | 12 months
  To compare the distribution profile of the daily physical activity (very sedentary, sedentary, moderately active) at 12 months between the intervention and control groups
Health-related quality of life | 12 months
  To evaluate the long-term effect of the health education program on the score of the COPD Assessment Test.
Rate of moderate or severe COPD exacerbations | 12 months
  To analyze the effect of the health education program on the risk and rate of moderate or severe COPD exacerbations
Relationship between change in physical activity level (PAL) and modification of health-related quality of life | 12 months
  To assess the relationship between the change of the PAL and the modification of the score of the CAT
Relationship between change in physical activity level (PAL) and exacerbations rate | 12 months
  To assess the relationship between the change of the PAL and rate of moderate or severe COPD exacerbations
Determinants of a clinically relevant increase of the physical activity level | 12 months
  To identify the determinants of a clinically relevant increase of the PAL (> 0.14 units) in patients with moderate-very severe COPD

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Garcia-Rio, MD, Study Chair — Hospital Universitario La Paz, IdiPAZ
Locations (1):
- Hospital Universitario La Paz-IdiPAZ, Madrid, Spain